CLINICAL TRIAL: NCT07294417
Title: Bone Cement Augmented Transpedicular Screw Fixation Versus Cannulated Screws Fixation in Osteoporotic Spine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Anas Zahra, Lecturer of Neurosurgery, Faculty of Medicine, KafrElsheikh University, KafrElsheikh, Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-824
Record Dates: First submitted 2025-12-06; First posted 2025-12-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Bone Cement Augmented Transpedicular Screw Fixation; Cannulated Screws Fixation; Osteoporotic Spine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients will be treated with bone cement augmented transpedicular screw fixation.
  Interventions: Procedure: Bone Cement Augmented Transpedicular Screw Fixation
- Group B (Active Comparator): Patients will be treated with cannulated pedicle screw fixation.
  Interventions: Procedure: Cannulated Screws Fixation

INTERVENTIONS:
Procedure: Bone Cement Augmented Transpedicular Screw Fixation — Patients will be treated with bone cement augmented transpedicular screw fixation.
  Arms: Group A
Procedure: Cannulated Screws Fixation — Patients will be treated with cannulated pedicle screw fixation.
  Arms: Group B

SUMMARY:
This study aims to compare the clinical and radiological outcomes of bone-cement-augmented transpedicular screw fixation versus cannulated pedicle screw fixation in patients with osteoporotic spines requiring posterior instrumentation, with respect to implant stability (loosening/pull-out), pain relief, functional recovery, and complication rates.

DETAILED DESCRIPTION:
Osteoporosis of the spine presents a significant challenge in spine surgery, particularly when instrumentation is needed for stabilization. With declining bone mineral density, conventional pedicle screw purchase becomes unreliable, leading to increased rates of screw loosening, pull-out, and fixation failure.

A relevant development in instrumentation has been the use of cannulated pedicle screws, sometimes in combination with cement-injectable systems, designed to allow cement to flow through the screw to reinforce fixation. Such systems have shown improved implant stability and lower failure rates in osteoporotic bone compared with solid screws.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Both sexes.
* Patients with confirmed osteoporosis on dual-energy X-ray absorptiometry (DEXA) scan (T-score ≤ -2.5),
* Patients presented with painful osteoporotic vertebral fractures, degenerative instability, or traumatic compression fractures.
* Patients are unresponsive to conservative management and require surgical stabilization.

Exclusion Criteria:

* Patients with healed or stable fractures respond to medical treatment.
* Patients with uncontrolled coagulopathy, active spinal infections such as discitis or osteomyelitis.
* Patients with spinal deformity exceeding thirty degrees, or vertebral body collapse greater than seventy percent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of wound infection | 6 months post-procedure
  Incidence of wound infection will be recorded.

SECONDARY OUTCOMES:
Incidence of complication rates | 6 months post-procedure
  Incidence of complication rates will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.